CLINICAL TRIAL: NCT01650831
Title: Clinical Study to Evaluate the Equivalence of the Modified BreathID Compared to Currently Approved BreathID System in Detection of H.Pylori Infection
Brief Title: Show Equivalence of the Modified BreathID Compared to Currently Approved BreathID in H.Pylori Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HP-MBI-0212
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Suspicion of Being Infected With H.Pylori
Keywords: Helicobacter Pylori; 13C Urea Breath Test; BreathID

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clinical Suspicion of Hpylori (Active Comparator): All subjects arriving at clinic with suspicion of having Helicobacter infection due to symptoms such as reflux, ulcer, gastric cancer and other clinical gastric conditions
  Interventions: Device: Modified BreathID

INTERVENTIONS:
Device: Modified BreathID — A new modified device, compared to the originally cleared BreathID measures breath from a subject via a nasal cannula
  Other Names: BreathID Hp

SUMMARY:
The purpose of this study is to confirm equivalence of a new generation breath analyzer (Modified BreathID) in its ability to detect H. pylori compared to the currently approved BreathID® System.

DETAILED DESCRIPTION:
The ¹³C-Urea Breath Test (UBT) is a non-invasive test for detecting the presence of Helicobacter pylori (H. pylori) infection by the organism's urease activity. In the presence of H. pylori, the ingestion of urea, labeled with the non-radioactive isotope 13C, results in production of labeled 13CO2, which can be quantified in expired breath. Each test is performed using a test kit consisting of a 13C-urea tablet and citrica powder to be dissolved in tap water ("13C-urea solution"). Before and after ingestion of the 13C-urea solution, samples of exhaled breath can be collected using a nasal cannula for real-time analysis and comparison to baseline concentrations. The patient's exhaled breath is analyzed and the ratio between 13CO2 and 12CO2 is computed. The patient is considered H. pylori positive when the difference between the ratios exceeds a predefined threshold (5 delta over baseline (DOB)). The current device marketed by Exalenz is large and costly. Exalenz has built a smaller, cheaper and more reliable new generation device for this application. Equivalence is being demonstrated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Present with clinical indication of H. pylori
3. Have the ability and willingness to sign the Informed Consent Form-

Exclusion Criteria:

1. Current serious disease
2. Participation in other trials
3. Antibiotics and/or Bismuth preparations for four (4) weeks prior to test
4. PPI or H2 blockers for two (2) weeks prior to test
5. Childbearing or breastfeeding women
6. Based on opinion of investigator, subject should not be enrolled in this trial
7. Allergy to citrus juice
8. Post -eradication therapy for H. pylori

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Liu, MD, Principal Investigator — Unimed Medical Center
Locations (1):
- Unimed Center, East Brunswick, New Jersey, United States

REFERENCES:
- [Background] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult subjects with suspected infection of Helicobacter Pylori due to symptoms were offered to do the test on a walk- in basis were recruited. 113 Subjects were recruited in October and November 2012 in a private medical clinic.
Pre-assignment Details: Subjects with prior knowledge of Helicobacter Pylori infection or taking proton pump inhibitors within the two week period before the test, were not included.Only one test per subject was done.
Groups:
- Clinical Suspicion of Hpylori: All subjects arriving at clinic with suspicion of having Helicobacter infection due to symptoms such as reflux, ulcer, gastric cancer and other clinical gastric conditions
  Modified BreathID : A new modified device, compared to the originally cleared BreathID measures breath from a subject via a nasal cannula
Period: Overall Study
Arm/Group | Clinical Suspicion of Hpylori
Started | 113
Completed | 112
Not Completed | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Suspicion of Hpylori
Number analyzed (Participants) | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (16.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Dichotomous (Presence/Absence of H.Pylori) Outcome Agreement in Diagnosis of H. Pylori
Description: The marketed (cleared) BreathID device and the investigational modified new generation BreathID device will measure simultaneously before (baseline) and after ingestion of substrate. The subject will be connected to both devices. The maximum time of measurement is 25 minutes.
Time Frame: 25 minutes
Population: Only subjects that had no recent knowledge of existing H.pylori infection and who met all protocol criteria and had no major protocol deviations, were included in the final analysis set (PP-per protocol).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clinical Suspicion of Hpylori
Number analyzed (Participants) | 79
Percentage of participants
  Positive agreeement | 100 [81.57 to 100]
  Negative agreement | 96.8 [88.98 to 99.11]

2. Primary Outcome: Positive/Negative for H.Pylori With Cleared BreathID
Description: The amount of subjects that produced positive/negative results with cleared BreathID device
Time Frame: 1 hour
Population: Per protocol positive/negative when testing with marketed BreathID
Measure: Number; unit: participants
Groups:
- Marketed BreathID Positive: Cleared BreathID subjects that were found to be positive for H.pylori
- Marketed BreathID Negative: Cleared BreathID subjects that were found to be negative for H.pylori
Arm/Group | Marketed BreathID Positive | Marketed BreathID Negative
Number analyzed (Participants) | 79 | 79
participants | 17 | 62

3. Primary Outcome: Positive/Negative for H.Pylori With Modified BreathID
Description: The amount of subjects that produced positive/negative results for H.pylori with modified BreathID
Time Frame: 1 hour
Population: Per protocol subjects tested with modified BreathID
Measure: Number; unit: participants
Groups:
- Positive Modified BreathID: The amount of subjects that produced positive results for H.pylori with modified BreathID.
- Negative Modified BreathID: The amount of subjects that produced negative results for H.pylori with modified BreathID.
Arm/Group | Positive Modified BreathID | Negative Modified BreathID
Number analyzed (Participants) | 79 | 79
participants | 19 | 60

ADVERSE EVENTS:
Arm/Group | Clinical Suspicion of Hpylori
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No